CLINICAL TRIAL: NCT03741816
Title: Randomized Blind Clinical Trial, Two-armed, Parallel of Indirect Pulp Capping With Biodentine and TheraCal LC in Permanent Mature Molars With Deep Carious Lesions
Brief Title: Indirect Pulp Capping With Biodentine and TheraCal LC in Permanent Mature Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Cristina Pasarín Linares, Teaching Assistant, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/2018
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Deep Carious Lesions; Reversible Pulpitis; Indirect Pulp Capping
Keywords: permanent molars; indirect pulp capping; reversible pulpitis; deep carious lesions; Biodentine; TheraCal LC

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine (Active Comparator): Indirect pulp capping with Biodentine in mature permanent molars with deep carious lesions and reversible pulpitis
  Interventions: Drug: Indirect pulp capping
- TheraCal LC (Experimental): Indirect pulp capping with TheraCal LC in mature permanent molars with deep carious lesions and reversible pulpitis
  Interventions: Drug: Indirect pulp capping

INTERVENTIONS:
Drug: Indirect pulp capping — Indirect pulp capping is a procedure in which a material is placed on a thin partition of remaining carious dentin that, if removed might expose the pulp.

SUMMARY:
Management of deep carious lesions in permanent mature molars with reversible pulpitis represents a challenge for clinicians. Vital pulp therapy includes indirect and direct pulp capping, partial pulpotomy and full pulpotomy. Indirect pulp capping is a procedure in which a material is placed on a thin layer of remaining soft dentin that, if removed, might expose the pulp. The objective is dentin bridge formation and pulp vitality preservation.

The aim of this randomized clinical trial is to evaluate the success rate of indirect pulp capping with Biodentine and TheraCal LC in mature permanent molars with deep carious lesions at one-year follow-up examination. The null hypothesis tested will be that there is no statistically significant difference in success rate between both materials in indirect pulp capping of permanent mature molars with deep carious lesions.

DETAILED DESCRIPTION:
Treatment options for permanent mature molars with deep carious lesions and a preoperative diagnosis of reversible pulpitis are varied among clinicians. In the last few years, a more biological approach is arising interest in the field of Endodontics through the development of calcium-silicate based cements that are used in vital pulp therapy.

A great variety of materials have been employed for indirect pulp capping. Although calcium hydroxide has been the "gold standard" for decades for this procedure, nowadays calcium-silicate based cements such as Mineral Trioxide Aggregate (MTA) are preferred. The second generation of these cements, among which Biodentine (Septodont, Saint Maur-des-Fossés, France) and TheraCal LC (Bisco, Schaumburg, IL, USA) stand out, try to overcome the first generation limitations.

On the other hand, there is a paradigm shift in caries removal techniques. Nowadays, the non-selective technique is not longer recommended and a selective removal technique until soft dentin is preferred in deep cavitated lesions.

The study will be carried out at the dental clinic of the Master of Restorative Dentistry and Endodontics (Medical and Dental School) of University of Valencia (Spain).

The study protocol that will be followed is:

1. Sample size estimation: 212 participants (106 per group).
2. Informed written consent will be obtained from all participants.
3. A full dental and medical history will be obtained from all patients.
4. Clinical (thermal and electric pulp tests, and palpation and percussion) and a radiographic examination (periapical radiograph and a small-volume cone beam computed tomography (CBCT).
5. Anesthesia administration and rubber dam placement.
6. Selective caries removal technique with high-speed diamond burs with air/water spray for enamel and Cariosolv gel and hand instruments until soft dentin.
7. Allocation to one of the two groups: Biodentine (control) or TheraCal LC (experimental) for indirect pulp capping procedures.
8. Final direct composite restoration using the selective etching technique and an universal adhesive.
9. Baseline periapical radiograph.
10. Follow-up: clinical and radiographic follow-up examinations will be conducted at one month, six months and twelve months (±2 weeks). In the one-year follow-up examination, a small-volume CBCT will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years without any systemic disease.
2. Presence of a deep carious lesion in a permanent mature molar without periapical pathology that penetrates radiographically into the inner dentin half or even third/ quarter.
3. Preoperative diagnosis of reversible pulpitis.
4. After selective caries removal to soft dentin with a high-speed diamond bur and Cariosolv gel and hand instruments, no pulpal exposure occurred.

Exclusion Criteria:

1. Negative response to pulp sensibility tests.
2. Clinical symptoms of irreversible pulpitis or pulp necrosis.
3. Presence of fistula, swelling, tenderness to percussion, tooth mobility.
4. Presence of periapical pathology on periapical radiographs (internal or external root resorption, abscence of normal appearance of periodontal ligament, presence of interradicular or periapical radiolucencies).
5. Pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
response to pulp sensibility testing ( thermal and electric pulp testing) | one year
  abscence of clinical signs and/or symptoms and radiographic findings of pulp degeneration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No